CLINICAL TRIAL: NCT06608888
Title: Unveiling the Neural Mechanisms of 5-HT7 in Sleep Apnea Induced by Arousal Dysregulation
Status: Recruiting | Type: Observational
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Principal Investigator, Jingying Ye, Chief Physician of Otorhinolaryngology, Beijing Tsinghua Changgung Hospital.Professor of Tsinghua Medicine, Tsinghua University., Beijing Tsinghua Chang Gung Hospital
Other Study IDs: 23657-0-01; 82341247 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2024-09-16; First posted 2024-09-23 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Arousal Dysregulation; Arousal Threshold; Lateral Hypothalamus; 5-HT7 Receptor
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-OSA patients group: Healthy individuals (without snoring symptoms, AHI < 5 events/h)；Simple snorers (with snoring symptoms, AHI < 5 events/h)
  Interventions: Diagnostic Test: MRI
- OSA patients: Patients diagnosed with OSA
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Multimodal MRI technology is a method that combines various magnetic resonance imaging techniques, providing more comprehensive images and information about human tissues and organs. These different imaging techniques include, but are not limited to:
  Structural MRI (sMRI): Provides information about the types of brain tissues, such as gray matter, white matter, and cerebrospinal fluid.
  Functional MRI (fMRI): Dynamically measures the hemodynamic response related to brain neural activity, commonly used to study brain functional activities.
  Diffusion Tensor Imaging (DTI): Offers information on the structural connections between brain regions, which can be used to study the neural fiber pathways of the brain
  Other Names: PSG; Genioglossus Electromyography

SUMMARY:
Obstructive sleep apnea (OSA), recognized as a highly prevalent sleep breathing disorder with severe complications, features a complex etiology. Poor understanding of disease pathogenesis limits the overall efficacy of interventions. Studies have found that upregulation of 5-HT7 expression in the lateral hypothalamus (LH) could reduce arousal threshold (ArTH) and induce an inhibitory effect to the respiratory central, which was associated with hypoxic stimulation. Therefore, the investigators speculate that the structural/functional abnormalities of the arousal-respiratory neural circuit, mediated by LH5-HT7, may play an important role in the pathogenesis of OSA. To verify the hypothesis, the investigators will compare the ArTH and the brain network presenting by multimodal MRI in normal individuals, snoring individuals, and OSA patients, to reveal the correlation between arousal dysregulation and the structure/function of LH regions; compare the changes of ArTH and brain network in OSA patients with low ArTH before and after CPAP treatment, to verify the interaction between hypoxia and arousal dysregulation, as well as whether the damaging performance of the arousal-respiratory brain regulation area in OSA patients can be partially reversed by relieving hypoxia. Above all, the joint application B team will further analyze the LH5-HT7 neural mechanism in the pathogenesis of OSA.

DETAILED DESCRIPTION:
The study consists of two parts: The first part is a cross-sectional study comparing the differences in arousal threshold, loop gain, and the brain network structure and functional connectivity of the brain areas involved in micro-arousal-respiratory center regulation between the non-OSA group (including healthy individuals and those with simple snoring) and the OSA group; The second part is a cohort study, which conducts a three-month longitudinal follow-up of the OSA group to observe the changes in the indicators of the structure and function of the core brain areas related to ArTH and micro-arousal-respiratory center regulation after the correction of intermittent hypoxia through CPAP treatment.The specific research content is as follows:

1. ArTH Comparative Analysis Based on Multimodal Assessment of OSA Etiology Select untreated OSA patients, simple snorers (with snoring symptoms, AHI < 5 events/h), and healthy individuals (without snoring symptoms, AHI < 5 events/h), matched for age and gender, and divide them into two groups.Non-OSA group (including healthy individuals and those with simple snoring) and OSA group . After all study participants have undergone upper airway CT, they are all subjected to overnight PSG with synchronous esophageal pressure monitoring, end-tidal carbon dioxide monitoring, and genioglossus electromyography (GGEMG) monitoring. A pharyngeal pressure regulation device is used to induce respiratory events with micro-arousals in the study participants under resistive ventilation, and the trends of ArTH, GGEMG, and respiratory drive (loop gain, LG) are analyzed among different sleep stages. Then, by integrating the above multimodal etiological parameters, the differences in micro-arousal regulation between OSA patients (high airway resistance and hypoxia group), simple snorers (high airway resistance without hypoxia group), and healthy individuals (low airway resistance without hypoxia group) are clarified. Furthermore, the weight of ArTH in the etiology of OSA is calculated, and the individual differences in ArTH among OSA patients and its correlation with the severity of the disease are analyzed.
2. Feature Analysis of OSA Micro-arousal-Respiratory Central Regulation Network Based on Multimodal MRI By integrating multimodal MRI imaging data, including structural T1, diffusion tensor imaging (DTI), and resting-state functional magnetic resonance imaging (rs-fMRI), the differences in brain network structure and functional connectivity of brain regions involved in micro-arousal-respiratory central regulation between OSA patients, simple snorers, and healthy individuals with different ArTH levels are compared. This reveals the patterns of functional connectivity changes and structural basis related to micro-arousal abnormal regulation in OSA patients, and clarifies the correlation with the lateral hypothalamus (LH) brain region.
3. Comparative Analysis of LH-Related Brain Region Structure and ArTH in OSA Patients with Low ArTH Before and After CPAP Treatment After OSA patients with different ArTH levels have undergone more than 6 months of CPAP treatment, ArTH and multimodal MRI imaging data (T1, DTI, rs-fMRI) are re-measured to observe the changes in ArTH and the structure/function of the core brain regions regulating micro-arousal-respiratory central in OSA patients after correcting intermittent hypoxia with CPAP treatment. These changes are compared with the ArTH and brain network structure of healthy controls to verify the damaging effects of hypoxia on brain networks and to clarify whether the damaging manifestations of the micro-arousal-respiratory central regulation regions in OSA patients can be partially reversed with treatment.

ELIGIBILITY:
Inclusion Criteria:

OSA Patients:

* Age between 20 and 60 years.
* Symptoms of sleep snoring and daytime sleepiness.
* Confirmed diagnosis of OSA following overnight sleep monitoring.

Simple Snorers:

* Age between 20 and 60 years.
* Symptoms of sleep snoring.
* Overnight sleep monitoring indicates not meeting the OSA diagnosis.

Healthy Controls:

* Age between 20 and 60 years.
* No symptoms of sleep snoring.
* Overnight sleep monitoring rules out the diagnosis of OSA.

Exclusion Criteria:

* Presence of severe pulmonary, neurological, or cardiovascular complications.
* History of long-term non-invasive positive pressure ventilation treatment (more than 3 months) or upper airway surgery.
* Sleep-disordered breathing due to special etiologies such as hypothyroidism, acromegaly, vocal cord paralysis, etc.
* Presence of severe mental illness, long-term alcohol abuse, or a history of prolonged use of sedative-hypnotic drugs.
* Central sleep apnea predominant sleep disorders due to various causes.
* Severe craniofacial deformities, myasthenia gravis, or other known myopathic histories.
* Patients with peripheral neuropathy caused by diabetes, autoimmune diseases, etc.
* Patients with comorbid insomnia, anxiety, depression, or other types of sleep disorders.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Snoring Population: Individuals who regularly experience snoring during sleep, often resulting in loud and disruptive noises.
  Healthy Volunteer Population: Individuals characterized by the absence of sleep disorders or other health conditions that could affect sleep quality. These volunteers typically exhibit regular sleep patterns without snoring or sleep-disordered breathing and meet specific age and health criteria to ensure they represent a healthy comparison group.
  OSA (Obstructive Sleep Apnea) Patient Population: Patients diagnosed with OSA, a sleep disorder where the airway collapses or becomes blocked repeatedly during sleep.OSA is typically confirmed through an overnight sleep study that measures breathing interruptions and oxygen desaturation events.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Arousal threshold | Three-month follow-up
  Calculate the patient's arousal threshold based on PSG results.
Fractional anisotropy | After three months of CPAP treatment, DTI were taken again on OSA patients to calculate the FA values.
  The fractional anisotropy (FA) value, obtained through diffusion tensor imaging (DTI) measurements, was used to compare the brain functions between patients with obstructive sleep apnea (OSA) and those without. Additionally, a follow-up was conducted after three months of continuous positive airway pressure (CPAP) treatment for OSA patients to compare the FA values before and after treatment, thereby clarifying the changes in patients' brain functions.
Connectivity strength | After three months of CPAP treatment, fMRI were taken again on OSA patients to calculate connectivity strength.
  The investigators conducted functional MRI measurements on patients with obstructive sleep apnea (OSA) and non-OSA volunteers, calculated functional connectivity, and compared the differences in their results. Subsequently, the investigators followed up with the OSA patients who underwent three months of CPAP therapy and compared the functional connectivity of brain regions before and after treatment to clarify changes in patients' brain functions.

SECONDARY OUTCOMES:
Sleep Stage Distribution | Three-month follow-up
  One of the indicators in PSG results.
Apnea-Hypopnea Index | Three-month follow-up
  One of the indicators in PSG results.
Oxygen Saturation | Three-month follow-up
  One of the indicators in PSG results.

CONTACTS AND LOCATIONS:
Overall Officials: Jingying Ye, Principal Investigator — BeijingTsinghua Changgung Hospital，Tsinghua University
Locations (1):
- No. 168 Litang Road, Changping District, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
all IPD that underlie results in a publication